CLINICAL TRIAL: NCT01773655
Title: Clinical and Histopathologic Characteristics of BAP1 Mutations
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 12-235
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Malignant Pleural Mesothelioma (MPM); Choroidal Nevus; Primary Uveal Melanoma (UM); Metastatic Uveal Melanoma (UM); Renal Cell Carcinoma; Cholangiocarcinoma
Keywords: somatic; germline; mutations; BAP1 (BRCA associated protein-1); 12-235
MeSH Terms: conditions — Mesothelioma, Malignant; Uveal Melanoma; Carcinoma, Renal Cell; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue specimens blood or saliva sample

GROUPS / COHORTS (1):
- tissue: This is a protocol to obtain and/or analyze tumor and germline DNA specimens of patients with MPM, choroidal nevus, and UM.
  Interventions: Other: tumor specimens

INTERVENTIONS:
Other: tumor specimens — All consenting patients (Consent 1) will participate in an anonymized assessment of the prevalence of germline BAP1 mutations. Available tumor specimens from patients with MPM and metastatic uveal melanoma will be tested for BAP1 mutation. Patients whose tumors harbor BAP1 mutations and/or meet the criteria for germline mutation specified in 2.2.2 will be approached for identified germline BAP1 testing after appropriate pre-test counseling (Consent 2).
  Patients who, through identified testing, are found to have germline BAP1 mutations will be asked to invite their relatives to participate in germline testing (Consent 3). First-degree relatives and any relatives with a malignancy will be prioritized. Expanding testing to family members of patients with BAP1 germline mutations is essential to delineate the penetrance and describe the various manifestations of this new cancer predisposition syndrome.

SUMMARY:
The goal of this protocol is to determine the prevalence of somatic and germline mutations in BAP1 (BRCA associated protein-1) among patients with mesothelioma , choroidal nevus, primary uveal melanoma (UM), or metastatic UM seen at our institution.

ELIGIBILITY:
Inclusion Criteria:

All consents:

* > or = to 18 years of age
* Ability to provide informed consent

Consent 1:

Mesothelioma

* Histologically proven diagnosis of Mesothelioma OR Choroidal nevus
* Diagnosis of choroidal nevus by direct examination and/or ultrasound/optical coherence tomography and possibly fluorescein angiography OR Primary uveal melanoma
* Diagnosis of uveal melanoma by direct examination and/or ultrasound/optical coherence tomography and possibly fluorescein angiography

Consent 2:

Mesothelioma

* Histologically proven diagnosis of Mesothelioma AND
* BAP1 mutation or loss of expression identified in tumor sample

OR one of the following:

* Age<50 at diagnosis
* No history of asbestos exposure
* Personal history of choroidal nevus, uveal melanoma, melanoma, renal cell carcinoma, or cholangiocarcinoma
* Family history of choroidal nevus, uveal melanoma, mesothelioma, renal cell carcinoma, or cholangiocarcinoma
* History of malignancy in more than two first-degree relatives OR Choroidal nevus
* Diagnosis of choroidal nevus by direct examination and/or ultrasound/optical coherence tomography and possibly fluorescein angiography AND one of the following:
* More than one clinical risk factor, which may include: orange pigment, thickness > 1 < 2.5mm
* Personal history of uveal melanoma, skin melanoma, mesothelioma renal cell carcinoma, or cholangiocarcinoma
* Family history of choroidal nevus, uveal melanoma, mesothelioma renal cell carcinoma, or cholangiocarcinoma OR Primary uveal melanoma
* Diagnosis of uveal melanoma by direct examination and/or ultrasound/optical coherence tomography and possibly fluorescein angiography

AND one of the following:

* Personal history of uveal melanoma, skin melanoma, mesothelioma, renal cell carcinoma, or cholangiocarcinoma
* Family history of choroidal nevus, uveal melanoma, mesothelioma, renal cell carcinoma, or cholangiocarcinoma
* History of malignancy in more than two first-degree relatives OR Metastatic uveal melanoma
* Histologically proven diagnosis of metastatic uveal melanoma AND
* BAP1 mutation or loss of expression identified in tumor sample

OR one of the following:

* Personal history of uveal melanoma, skin melanoma, mesothelioma renal cell carcinoma, or cholangiocarcinoma
* Family history of choroidal nevus, uveal melanoma, mesothelioma renal cell carcinoma, or cholangiocarcinoma
* History of malignancy in more than two first-degree relatives

Consent 3:

* Relative of patient with germline BAP1 mutation identified through identified testing

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC's clinics
Sampling Method: Non-Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2013-01; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
determine the prevalence of germline BAP1 mutations | 2 years
  Prevalence will be estimated as the proportion of all specimens who tested positive for mutation, and reported along with the corresponding exact 95% confidence intervals.

SECONDARY OUTCOMES:
prevalence of somatic BAP1 mutations in disease mesothelioma and metastatic uveal melanoma. | 2 years
  The frequency of somatic mutations will be tabulated by factors of interest such as:
  * personal and familial risk factors: age, smoking, and asbestos mesothelioma, personal and family history of cancer or of related diseases (mesothelioma and metastatic uveal melanoma)
  * disease characteristics: histology, stage, location, site of metastasis (if present) (for mesothelioma and metastatic uveal melanoma); COMS criteria, GEP class, number of clinical risk factors (for metastatic uveal melanoma)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Zauderer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT01773655/ICF_000.pdf